CLINICAL TRIAL: NCT05375851
Title: Digital Interventions As an Add-on Tool in Generalized Anxiety Disorder Treatment: a Randomized Clinical Trial
Brief Title: Digital Interventions As an Add-on Tool in Generalized Anxiety Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54357621.7.0000.5327
Record Dates: First submitted 2022-04-14; First posted 2022-05-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: digital mental health; mobile applications; measurement-based care; GAD-7; psychoeducation; generalized anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As we are going to use a digital tool as an adjunct to the treatment and as the clinician also needs to guide the patient during this intervention and discuss with him about the content of the videos and the results of the scales, there is no possibility of blinding these parts, however, we opted for blind the evaluator who will carry out the baseline, mid-term and end-of-study evaluations. The study coordinator will talk to each patient to advise them not to reveal which group they participated during the interview with the blinded evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Intervention (Experimental): The digital interventions will consist of two parts:
  A) Psychoeducation videos: Five psychoeducation videos on mental health and GAD will be produced especially for the research to be watched by the patient between consultations. These videos will last approximately 3 minutes, will use animations and educational content. They will be available on "+PSI" app. The topics of the videos will be as follows: Normal Anxiety versus Pathological Anxiety; Sleep Hygiene; Healthy Eating and Mental Health; Physical Exercise and Mental Health; Excessive Consumption of Alcohol and Drugs.
  B) GAD-7 Scale: The patient will be instructed to respond to the GAD-7 self-administered scale the day before their next scheduled appointment. This instrument will also be available free of charge on +PSI mobile app and will be used to guide clinical management.
  The above digital interventions will be added to the usual GAD treatment.
  Interventions: Other: Digital Interventions; Drug: Treatment as Usual
- Control (Active Comparator): The usual treatment will be standardized as follows:
  Biweekly online consultations (via WhatsApp or Google Meet) previously scheduled, 20/30 minutes-long, with a trained psychiatrist.
  The patient will receive only clinical, not psychotherapeutic treatment. The psychiatrist will be instructed to perform an assessment of symptoms, general guidelines on the pathology, use of medication when necessary.
  The medication of choice, when necessary, will be fluoxetine, as it is the medication for the treatment of GAD available free of charge in our health system in Brazil.
  Interventions: Drug: Treatment as Usual

INTERVENTIONS:
Other: Digital Interventions — The digital interventions will consist of two parts:
  A) Psychoeducation videos: Five psychoeducation videos on mental health and GAD will be produced especially for the research to be watched by the patient between consultations. These videos will last approximately 3 minutes, will use animations and educational content. They will be available on "+PSI" app. The topics of the videos will be as follows: Normal Anxiety versus Pathological Anxiety; Sleep Hygiene; Healthy Eating and Mental Health; Physical Exercise and Mental Health; Excessive Consumption of Alcohol and Drugs.
  B) GAD-7 Scale: The patient will be instructed to respond to the GAD-7 self-administered scale the day before their next scheduled appointment. This instrument will also be available free of charge on +PSI mobile app and will be used to guide clinical management.
  Arms: Digital Intervention
Drug: Treatment as Usual — The usual treatment will be standardized as follows:
  Biweekly online consultations (via WhatsApp or Google Meet) previously scheduled, 20/30 minutes-long, with a trained psychiatrist.
  The patient will receive only clinical, not psychotherapeutic treatment. The psychiatrist will be instructed to perform an assessment of symptoms, general guidelines on the pathology, use of medication when necessary.
  The medication of choice, when necessary, will be fluoxetine, as it is the medication for the treatment of GAD available free of charge in our health system in Brazil.
  Other Names: Care as Usual

SUMMARY:
Background: Over the last several years, there has been an increase in the popularity and availability of mobile digital technologies. Many recent studies have evaluated a range of mobile digital mental health interventions (DMHIs). Smartphone applications, remote monitoring, tracking devices, and wearable computers such as smartwatches and virtual reality headsets are being widely used for these studies. Besides that, psychometric scales are being used to help psychiatrists to improve treatment outcomes. The systematic administration of symptom rating scales and other assessment tools to help treatment decisions has been called measurement-based care (MBC) and it has shown good results in improving outcomes and time to response/remission of psychiatric diseases. As there is little data regarding MBC in Generalized Anxiety Disorder (GAD), the investigators decided to put technology and MBC together to study an easy and accessible way to improve the GAD usual treatment. Objectives: The aim of this study is to evaluate the benefit of digital interventions as an add-on tool to "treatment-as-usual" (TAU) in GAD patients. Methods: A twelve-weeks randomized clinical trial will be performed with 60 GAD patients. The control group will receive TAU, defined as 30-minutes online consultation with a trained psychiatrist, consisting in symptoms evaluation, general orientations about the disorder and use of medication. The consultations are going to occur biweekly. The digital intervention group (active group) will receive TAU, associated with two digital tools. The first one consists of psychoeducational videos to be seen between the sessions and the second one includes self-application of GAD-7 scale the day before the next scheduled consultation. All these digital interventions are going to be accessed in a mobile application, called "+PSI", that is already available in Apple Store and Google Play. The participants are going to be instructed to download the application on their mobile phones for free. The videos are going to be created especially for this project and will use animations and educational content, being of short duration (average 3 minutes). GAD-7 scale, and Hamilton Anxiety Scale (HAM-A) are going to be applied at baseline and at the end of the follow up by a blind rater. The investigators are also going to test the application tools usability using the System Usability Scale (SUS). Intermediate and follow-up evaluations will be performed to assess the speed and maintenance of improvement, respectively.

DETAILED DESCRIPTION:
* This study will follow the CONSORT guideline as a guide for conducting a clinical trial.
* The sample size was calculated to detect differences in the mean variation in the GAD-7 score (difference between the initial GAD-7 and the final GAD-7) between the Digital Intervention and Control Groups, with a difference of 5 points as relevant for the study. For this, the PSS Health tool version 0.1.6 was used. Considering a power of 80%, a significance level of 5% and a standard deviation of 6 points, the total sample size was 46 subjects, 23 in each group. Adding 30% for possible losses and refusals, the sample size should be 60 (30 in each group).
* Statistical analysis will be performed using descriptive statistics (mean, mode, median, standard deviation, frequencies and percentages). Student's t test will be used to compare means of independent variables. In the conclusions of the statistical tests, a significance level of 5% will be used, that is, whenever p < 0.05 there is evidence of statistical significance.
* The analyzes are going to use intention-to-treat model, preserving the benefit of randomization and avoiding biases due to exclusion and/or loss of patients during the research.
* The digital interventions will consist of two parts:

A) Psychoeducation videos: Five psychoeducation videos on mental health and GAD will be produced especially for the research to be watched by the patient between consultations. These videos will last approximately 3 minutes, will use animations and educational content. They will be available free of charge for the patient to watch on Artmed's "+PSI" app, available on both the Apple Store and Google Play. The topics of the videos will be as follows: Normal Anxiety versus Pathological Anxiety; Sleep Hygiene; Healthy Eating and Mental Health; Physical Exercise and Mental Health; Excessive Consumption of Alcohol and Drugs.

B) GAD-7 Scale: The patient will be instructed to respond to the GAD-7 self-administered scale the day before their next scheduled appointment. This instrument will also be available free of charge on Artmed's +PSI mobile application and will be used to guide clinical management.

* The usual treatment will be standardized as follows:

  * Biweekly online consultations (via WhatsApp or Google Meet) previously scheduled, 20/30 minutes-long, with a trained psychiatrist.
  * The patient will receive only clinical, not psychotherapeutic treatment.
  * The psychiatrist will be instructed to perform an assessment of symptoms, general guidelines on the pathology, use of medication when necessary.
  * The medication of choice, when necessary, will be fluoxetine, as it is the medication for the treatment of GAD available free of charge in our health system in Brazil.
* The clinician may also opt for some other class of medication associated with the use of fluoxetine, such as benzodiazepines, for example, which must be duly recorded in the database (drug, dose, time of use). If the patient does not have an indication for the use of fluoxetine or does not tolerate its use, he will be excluded from the study and referred to the health unit in his region to evaluate other therapeutic possibilities.
* The follow-up of patients during the research protocol will occur biweekly, online. The videocalls will not be recorded. The duration of the study will be 12 weeks; each patient will have 6 consultations with their clinician.
* Always at the first appointment, the professional will indicate to the patient to download the application on his device (mobile or tablet) and will help him with technical questions. In the intervention group, the patient will leave the consultation with the indication and combination of homework. A video will be indicated to be watched before the next appointment, which will be discussed with the psychiatrist during the next session, debating the topic and clearing up possible doubts. It will also be arranged with the patient to complete the GAD-7 self-administered questionnaire the day before the next scheduled appointment. The result of this assessment will be shared with the practitioner in the next session, and both will discuss and evaluate the results together. If the patient in the intervention group has not seen the video or completed the scale as instructed before the scheduled time, the psychiatrist will do these activities with the patient during consultation time to ensure that he or she has exposure to the intervention.
* Always at the first appointment, the professional will indicate to the patient to download the application on his device (mobile or tablet) and will help him with technical questions. In the intervention group, the patient will leave the consultation with the indication and combination of homework. A video will be indicated to be watched before the next appointment, which will be discussed with the psychiatrist during the next session, debating the topic and clearing up possible doubts. It will also be arranged with the patient to complete the GAD-7 self-administered questionnaire the day before the next scheduled appointment. The result of this assessment will be shared with the practitioner in the next session, and both will discuss and evaluate the results together. If the patient in the intervention group has not seen the video or completed the scale as instructed before the scheduled time, the psychiatrist will do these activities with the patient during consultation time to ensure that he or she has exposure to the intervention.
* Between appointments 3 and 4, patients from both groups will be contacted by one of the blinded evaluators to perform the HAM-A. The purpose of applying this scale in the middle of the study is to assess whether there is a difference in response time between the digital intervention group and the control group.
* Patients will be re-contacted at 3 and 6 months after the end of the survey to complete the GAD-7 and HAM-A scales again, to assess long-term response maintenance and adherence to treatment.
* The Net Promoter scale will be used at the endpoint of the study to assess whether there was a difference in satisfaction with the received treatment between the control and intervention groups.
* As the investigators are going to use a digital tool as an adjunct to the treatment and as the clinician also needs to guide the patient during this intervention and discuss with him about the content of the videos and the results of the scales, there is no possibility of blinding these parts, however, the research group opted for blind the evaluator who will carry out the baseline, mid-term and end-of-study evaluations. The study coordinator will talk to each patient to advise them not to reveal which group they participated during the interview with the blinded evaluator.
* The investigators will also control by sex, age, socioeconomic class to understand whether digital tools can have a different impact on each group. The evaluation of the impact of psychiatric comorbidities will also be evaluated, analyzing them as confounders (presence of associated depression, for example).
* Adherence to the medication prescription will be controlled by counting pills at each visit together with the patient, to avoid confusion bias regarding the use or not of the medication correctly and the improvement of the patient. At each appointment, the patient will be guided by the attending physician to separate the exact number of pills until the date of the next appointment, when the number of remaining pills will be checked again, and the data duly recorded in the database.
* The research group will be composed of 12 members, duly trained for their distinct functions.
* After the selection of the team of professionals who will collaborate with the project, an online course will be given by the project coordinator with all members to explain the research protocol and training of all stages of the project, as well as regarding the evaluation instruments that will be used.
* During the entire course of the research, the assistant clinician will be aware of risks that patients may present during the study, such as suicide risk, for example. When such a situation is identified, the participant will be automatically disconnected from the study and will be referred to specific treatment for his/her condition (in case of suicide risk, the standard measures for this psychiatric emergency will be carried out and the patient will be referred to the nearest psychiatric emergency).
* The prescribed medication will be sent by email to the patient through the system for special prescriptions of the Regional Council of Medicine (CREMERS) and he will look for a Primary Care Center to take the medication. At the endpoint of the study, all patients will be referred to follow treatment in the basic health network closest to their residence, also considering that the medication used is already the medication that is available free of charge in Brazil's health system.
* The database will use RedCap resources, to which all members of this study will have access, always taking into account the necessary ethical precautions.
* All data added to the database will be reviewed by the research assistants daily. Any inconsistency will be immediately reported to the research coordinator.
* All participants will be invited to read, understand the research objectives, through the informed consent form before participating in the study. There is the possibility for the participant to withdraw from the study at any time.
* All data will be kept in a safe place by those responsible for the project, guaranteeing the privacy rights of the interviewees. Only team members will have access to and handle the data collected. Items referring to the confidentiality of the information collected will be guaranteed by the non-identification of subjects.
* The investigators expect that intervention group can show a greater clinical improvement in the assessment of the variation of initial and final GAD symptoms (baseline and endpoint delta), evaluated by GAD-7 and HAM-A scales. To be considered relevant in care practice, the expectation is that this improvement has both statistical and clinical significance.
* Another expected result is to find is that control group presents a higher dropout rate than intervention group, considering the hypothesis that the interventions associated with usual care that will be implemented add benefits of therapeutic bond and adherence to treatment. Furthermore, the investigators assume that the intervention group can start the improvement process faster than the control group and that this improvement will be sustained for longer (follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* diagnosis of GAD confirmed through MINI.
* access to internet and smartphone (or tablet with internet).

Exclusion Criteria:

* psychiatric comorbidities more severe than GAD (assessed using CGI).
* suicide risk.
* pregnancy or lactation.
* being in psychological/psychiatric treatment or having been in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical change as measured by the Generalized Anxiety Disorder-7 (GAD-7) scale score | The initial evaluation will take place before session 1 by a blinded evaluator and the final evaluation will take place shortly after the last session (12 weeks of treatment) also by a blinded evaluator.
  Patients will be evaluated at the beginning and at the endpoint of the study with the self-administered GAD-7 scale, and the difference found between the deltas (end minus initial) of the control and intervention groups will be considered the primary outcome of the study. The GAD-7 scale score ranges from 0 to 21 points. A score between 5 and 9 points characterizes mild GAD. Between 10 and 14, moderate GAD and between 15 and 21, severe GAD.

SECONDARY OUTCOMES:
Clinical improvement measured through Hamilton Anxiety (HAM-A) scale scores | The initial evaluation will take place before session 1 by a blinded evaluator and the final evaluation will take place shortly after the last session (12 weeks of treatment) also by a blinded evaluator.
  Patients will be evaluated at the beginning and at the endpoint of the study with HAM-A scale, and the difference found between the deltas (end minus initial) of the control and intervention groups will be considered a secondary outcome of the study. The HAM-A's total score ranges from 0 to 56. The higher the score, the greater the patient's degree of anxiety.
Treatment dropout rates | Session 1 until session 6 (12 weeks long)
  We will check if there was a significant difference between the dropout rates between the groups.
Speed of improvement measured by Hamilton Anxiety Scale (HAM-A) | Between 4 and 6 weeks after the start of the study (between session 3 and session 4)
  Patients will be evaluated if there was a difference in the speed of improvement between the groups. HAM-A is going to be applied between session 3 and 4 to check this difference. The HAM-A's total score ranges from 0 to 56. The higher the score, the greater the patient's degree of anxiety.
System usability evaluation | SUS will be applied through study completion, an average of 12 weeks after session 1
  We will use the System Usability Scale (SUS) to assess the usability of the system used to deliver the interventions. The SUS score varies from 0 to 100 points, with 0 representing the worst acceptance and 100 the best acceptance of the analyzed digital tool.
Level of satisfaction with the treatment received | NPS will be applied through study completion, an average of 12 weeks after session 1
  We will use the Net Promoter Scale (NPS) to assess the level of satisfaction with the treatment received. The NPS consists of a numerical and visual scale (with representative "emojis") ranging from 0 to 10 points, with 0 being the lowest level of satisfaction with the treatment received and 10 the highest level of satisfaction with the treatment received.
Relapse and treatment dropout rates after 3 and 6 months measured with Generalized Anxiety Disorder -7 scale (GAD-7) | 3 and 6 months after the end of the study
  Patients will be re-contacted at 3 and 6 months after the end of the study to complete GAD-7 scale. The GAD-7 scale score ranges from 0 to 21 points. A score between 5 and 9 points characterizes mild GAD. Between 10 and 14, moderate GAD and between 15 and 21, severe GAD.
Relapse and treatment dropout rates after 3 and 6 months measured with Hamilton Anxiety Scale (HAM-A) | 3 and 6 months after the end of the study
  Patients will be re-contacted at 3 and 6 months after the end of the study to complete HAM-A scale. The total score of HAM-A scale ranges from 0 to 56. The higher the score, the greater the patient's degree of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gisele G Manfro, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soobiah C, Cooper M, Kishimoto V, Bhatia RS, Scott T, Maloney S, Larsen D, Wijeysundera HC, Zelmer J, Gray CS, Desveaux L. Identifying optimal frameworks to implement or evaluate digital health interventions: a scoping review protocol. BMJ Open. 2020 Aug 13;10(8):e037643. doi: 10.1136/bmjopen-2020-037643. PMID 32792444
- [Background] Borghouts J, Eikey E, Mark G, De Leon C, Schueller SM, Schneider M, Stadnick N, Zheng K, Mukamel D, Sorkin DH. Barriers to and Facilitators of User Engagement With Digital Mental Health Interventions: Systematic Review. J Med Internet Res. 2021 Mar 24;23(3):e24387. doi: 10.2196/24387. PMID 33759801
- [Background] Graham AK, Lattie EG, Powell BJ, Lyon AR, Smith JD, Schueller SM, Stadnick NA, Brown CH, Mohr DC. Implementation strategies for digital mental health interventions in health care settings. Am Psychol. 2020 Nov;75(8):1080-1092. doi: 10.1037/amp0000686. PMID 33252946
- [Background] Stirman SW, Gutner CA, Langdon K, Graham JR. Bridging the Gap Between Research and Practice in Mental Health Service Settings: An Overview of Developments in Implementation Theory and Research. Behav Ther. 2016 Nov;47(6):920-936. doi: 10.1016/j.beth.2015.12.001. Epub 2015 Dec 21. PMID 27993341
- [Background] Schueller SM, Torous J. Scaling evidence-based treatments through digital mental health. Am Psychol. 2020 Nov;75(8):1093-1104. doi: 10.1037/amp0000654. PMID 33252947
- [Background] Firth J, Torous J, Nicholas J, Carney R, Rosenbaum S, Sarris J. Can smartphone mental health interventions reduce symptoms of anxiety? A meta-analysis of randomized controlled trials. J Affect Disord. 2017 Aug 15;218:15-22. doi: 10.1016/j.jad.2017.04.046. Epub 2017 Apr 25. PMID 28456072
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Background] Guo T, Xiang YT, Xiao L, Hu CQ, Chiu HF, Ungvari GS, Correll CU, Lai KY, Feng L, Geng Y, Feng Y, Wang G. Measurement-Based Care Versus Standard Care for Major Depression: A Randomized Controlled Trial With Blind Raters. Am J Psychiatry. 2015 Oct;172(10):1004-13. doi: 10.1176/appi.ajp.2015.14050652. Epub 2015 Aug 28. PMID 26315978
- [Background] Shaygan M, Yazdani Z, Valibeygi A. The effect of online multimedia psychoeducational interventions on the resilience and perceived stress of hospitalized patients with COVID-19: a pilot cluster randomized parallel-controlled trial. BMC Psychiatry. 2021 Feb 11;21(1):93. doi: 10.1186/s12888-021-03085-6. PMID 33573631
- [Background] Ghanbari E, Yektatalab S, Mehrabi M. Effects of Psychoeducational Interventions Using Mobile Apps and Mobile-Based Online Group Discussions on Anxiety and Self-Esteem in Women With Breast Cancer: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 18;9(5):e19262. doi: 10.2196/19262. PMID 34003138
- [Background] Fusar-Poli P, Correll CU, Arango C, Berk M, Patel V, Ioannidis JPA. Preventive psychiatry: a blueprint for improving the mental health of young people. World Psychiatry. 2021 Jun;20(2):200-221. doi: 10.1002/wps.20869. PMID 34002494
- [Background] Powell LA, Parker J, Weighall A, Harpin V. Psychoeducation Intervention Effectiveness to Improve Social Skills in Young People with ADHD: A Meta-Analysis. J Atten Disord. 2022 Feb;26(3):340-357. doi: 10.1177/1087054721997553. Epub 2021 Mar 5. PMID 33666104
- [Background] Rigabert A, Motrico E, Moreno-Peral P, Resurreccion DM, Conejo-Ceron S, Cuijpers P, Martin-Gomez C, Lopez-Del-Hoyo Y, Bellon JA. Effectiveness of online psychological and psychoeducational interventions to prevent depression: Systematic review and meta-analysis of randomized controlled trials. Clin Psychol Rev. 2020 Dec;82:101931. doi: 10.1016/j.cpr.2020.101931. Epub 2020 Oct 24. PMID 33137611
- [Background] Kessler RC, Angermeyer M, Anthony JC, DE Graaf R, Demyttenaere K, Gasquet I, DE Girolamo G, Gluzman S, Gureje O, Haro JM, Kawakami N, Karam A, Levinson D, Medina Mora ME, Oakley Browne MA, Posada-Villa J, Stein DJ, Adley Tsang CH, Aguilar-Gaxiola S, Alonso J, Lee S, Heeringa S, Pennell BE, Berglund P, Gruber MJ, Petukhova M, Chatterji S, Ustun TB. Lifetime prevalence and age-of-onset distributions of mental disorders in the World Health Organization's World Mental Health Survey Initiative. World Psychiatry. 2007 Oct;6(3):168-76. PMID 18188442
- [Background] Slee A, Nazareth I, Bondaronek P, Liu Y, Cheng Z, Freemantle N. Pharmacological treatments for generalised anxiety disorder: a systematic review and network meta-analysis. Lancet. 2019 Feb 23;393(10173):768-777. doi: 10.1016/S0140-6736(18)31793-8. Epub 2019 Jan 31. PMID 30712879
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shear MK, Vander Bilt J, Rucci P, Endicott J, Lydiard B, Otto MW, Pollack MH, Chandler L, Williams J, Ali A, Frank DM. Reliability and validity of a structured interview guide for the Hamilton Anxiety Rating Scale (SIGH-A). Depress Anxiety. 2001;13(4):166-78. PMID 11413563
- [Background] Wilberforce M, Poll S, Langham H, Worden A, Challis D. Measuring the patient experience in community mental health services for older people: A study of the Net Promoter Score using the Friends and Family Test in England. Int J Geriatr Psychiatry. 2019 Jan;34(1):31-37. doi: 10.1002/gps.4978. Epub 2018 Sep 24. PMID 30247775